CLINICAL TRIAL: NCT02629536
Title: Effect on Migraine Frequency of Combined Anti-oxidant Therapy: N-acetylcysteine, Vitamin E and Vitamin C (NEC): The MIGRANT Study
Brief Title: Effect on Migraine Frequency of Combined Anti-oxidant Therapy: The MIGRANT Study.
Acronym: MIGRANT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Notre Dame Australia (Other)
Responsible Party: Principal Investigator, Professor Eric Visser, Professor Eric J Visser, University of Notre Dame Australia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Churack Chair
Record Dates: First submitted 2015-12-03; First posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Migraine, Headaches
MeSH Terms: conditions — Migraine Disorders | interventions — Acetylcysteine; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active-verum-NAC tablet (Experimental): Intervention: Twice-daily administration of N-acetyl cysteine 600 mg, VitE 250 IU, VitC 500 mg tablets
  Interventions: Drug: N-acetyl cysteine 600 mg, VitE 250 IU, VitC 500 mg tablet
- Sham-placebo tablet (Placebo Comparator): Intervention: Twice daily administration of sham/placebo tablet
  Interventions: Drug: N-acetyl cysteine 600 mg, VitE 250 IU, VitC 500 mg tablet

INTERVENTIONS:
Drug: N-acetyl cysteine 600 mg, VitE 250 IU, VitC 500 mg tablet — N-acetyl cysteine 600 mg, VitE 250 IU, VitC 500 mg tablet
  Other Names: NEC

SUMMARY:
Migraine affects 15% of Western Australians and is a leading cause of suffering and disability in our community (1,2). Research suggests that inflammation of the brain's coverings (meninges) by nerve cell inflammation and the release of 'free radicals', is a cause of migraine. N-acetylcysteine, Vitamin E and Vitamin C are powerful anti-oxidants (free-radical scavengers) that reduce brain inflammation and nerve activity. It is therefore possible these anti-oxidants could reduce the number and severity of migraines. We will study 90 subjects to see if a combination of N-acetylcysteine 600 mg, Vitamin E 250 IU and vitamin C 500 mg (NEC) taken twice daily for 3 months, will reduce migraine attacks. This safe vitamin-based therapy has never been studied and if effective, will play an important role in migraine prevention.

DETAILED DESCRIPTION:
Summary:

Migraine affects 15% of Western Australians and is a leading cause of suffering and disability in our community. Research suggests that inflammation of the brain's coverings (meninges) by nerve cell inflammation and the release of 'free radicals', is a cause of migraine. N-acetylcysteine, Vitamin E and Vitamin C are powerful anti-oxidants (free-radical scavengers) that reduce brain inflammation and nerve activity. It is therefore possible these anti-oxidants could reduce the number and severity of migraines. We will study 90 subjects to see if a combination of N-acetylcysteine 600 mg, Vitamin E 250 IU and vitamin C 500 mg (NEC) taken twice daily for 3 months, will reduce migraine attacks. This safe vitamin-based therapy has never been studied and if effective, will play an important role in migraine prevention.

Because migraine is a complex neuro-vascular-inflammatory disorder with a 'cascade' of steps, there are many potentially targets for drug prophylaxis. Research highlights the importance brain neuro-inflammation mediated by Calcitonin Gene Related Peptide (CGRP) and Substance P (SP), and oxygen and nitrogen free radical species (FRS) (eg. nitric oxide [NO]) in the pathogenesis of migraine. Increased levels of NO and CGRP were found in the jugular venous blood migraineurs and NO produces cerebral vasodilation, which is a key step in migraine generation. Furthermore, FRS activate the trigeminal-cervical nucleus (TCN) which is the main centre of nociceptive (pain) sensitization in headaches-Sumatriptan blocks this process accounting for some of its anti-migraine effect.

Anti-oxidants such as N-acetylcysteine (NAc), Vitamin C (ascorbic acid) (VitC) and Vitamin E (alpha-tocopherol) (VitE) are potent FRS 'scavengers', which means they could be used to prevent migraine. Two small non-randomised trials suggested that antioxidants reduced migraine frequency and disability. Like sumatriptan, NAc reduces activation of the TCN by NO, also neuro-inflammation in brain disorders such as Parkinson's disease. VitC and VitE reduced NO levels in mice and VitC enhanced the neuro-inhibitory effects of gamma amino butyric acid in the central nervous system-This mechanism could conceivably interrupt 'spreading cortical activation' which is the first step in the migraine cascade.

Migraineurs have an increased risk of developing an analogous neuro-inflammatory disorder, Complex Regional Pain Syndrome (CRPS); increased plasma levels of SP, CGRP and FRS were found in patients with these conditions. CRPS responds to treatment with NAc and VitC. A meta-analysis found that combined (but not single-agent) anti-oxidant therapy (CAT) was safe and effective in treating chronic pancreatitis, an inflammatory pain disorder similar to both CRPS and migraine.

We previously proposed that migraine be considered a form of 'CRPS of the brain' which therefore (like CRPS) may also respond to CAT. Literature review confirmed this theory has not yet been explored. We will therefore test the hypothesis that twice-daily administration of a combination of NAC 600 mg, VitE 250 IU and VitC 500 mg (NEC) for 12 weeks, will significantly reduce migraine frequency. If proven effective, NEC will be an inexpensive, accessible and safe treatment for managing the burden of migraine in the Western Australian community

Experimental hypothesis Twice-daily administration of NEC (NAc 600 mg, VitE 250 IU and VitC 500 mg) for 12 weeks significantly reduces migraine frequency in patients who experience two-to-eight migraines per month, compared with a placebo-control group.

Methods: Study design is based on guidelines for migraine clinical trials of the International Headache Society (IHS) 2013. It will be a clinically-pragmatic, proof-of-concept investigation.

Trial design: Prospective, randomised, double-blind, placebo-controlled, two parallel-group trial.

Subjects: Males and females from 18 to 65 years of age.

Recruitment: Convenience sample of migraine patients attending general practice clinics, neurology clinics linked to UNDA Sydney and pain clinics (Joondalup Health Campus); via Headache Australia, Chronic Pain Australia, UNDA and Fremantle Hospital Research Foundation websites, and newspaper advertising, as required.

NB: Subjects stabilised on one migraine prevention drug were not excluded from the study, because cessation and washout of drugs would hinder recruitment and retention and does not reflect 'real-life' clinical practice.

Power calculation The population for an adequately powered RCT was calculated from data of similar studies in migraine prevention (30-35). It is estimated that 60% of subjects in the active study group and 30% in the placebo-control group will report a 'positive outcome' (≥ 30% reduction in headache frequency, from baseline). With 80% power and p<0.05, the study population for this RCT is 84 subjects. An interim proof-of-concept (pilot) analysis will be performed when 40 subjects (20 in each group) complete the study, based on guidelines for pilot studies by Lancaster et al.

Number of subjects: 84 subjects in total, 42 in each study group. Active study group (n=42) and placebo-control group (n=42).

Randomisation and blinding: Computer randomization of subjects will be in 'blocks' of 10, as per IHS migraine trial guidelines. Subjects, researchers and data analysts will be blinded. A pharmacist will dispense active (NEC) and sham trial drugs and maintain records.

Study duration: 16 weeks (112 days, or four months) total; four weeks baseline study phase (for stabilization and baseline measurements); 12 weeks active study phase. Start: January 1, 2016. Finish: January 1, 2017.

Study logistics and flow:

* Ethics approval.
* Advertising.
* Serial recruitment of subjects.
* Informed consent obtained.
* Study enrolment interview with a researcher.
* Subjects provided with a paper headache diary which they must complete a minimum of five days per week for 16 weeks of the study; should take no longer than 5 minutes per day.
* Four weeks baseline study phase, baseline outcomes measures.
* After baseline phase, subjects stratified as having < 3 ≥ migraines per month, as per IHS guidelines.
* Computer randomisation within these strata in 'blocks' of 10, as per IHS 2013.
* Randomised to active (NEC) or placebo-controlled (sham) study groups.
* They will need to take either verum or placebo tablet twice daily for 12 weeks.
* 12 week active study phase begins.
* Daily entries in headache diary.
* Control and compliance visits or phone contact every 4 weeks.
* Study termination face-to-face interview at the end of week 12.
* Collect diaries and left-over trial drugs.
* Data collated by blinded researcher.
* Statistical analysis performed by independent statistician.
* Data retained in a secure location for five years.

Data collection and analysis: Headache diary is based on; Headache diary-preventive therapies, versions 4, IHS guidelines for controlled trials of drugs in migraine, 2011. Headache diary must be completed for at least five days each week during the baseline and active study phases. Study drugs must be consumed on at least five days each week during the active study phase.

Intention-to-treat analysis: data from drop-outs and partial study completions will be analysed and reported.

Statistical analysis: Analysis by an independent, blinded biostatistician from the UNDA School of Medicine Health Research Institute, Fremantle WA, using SAS® version 9.2 statistical software (Cary NC, USA) and Excel spreadsheet 2007™ (Redmond WA, USA) statistical packages. Analysis of outcomes will be performed on the intention-to-treat population. Some post hoc analysis of data may be performed. Significance level: p<0.05; confidence limits of 95%.

Data sets: Demographic, clinical, outcomes data. Descriptive data: Frequencies, percentages (categorical data); means, standard deviations, confidence intervals (continuous data).

Comparative data analysis: Student's t test for continuous data; Chi square test for categorical data; confidence intervals; linear or logistic regression.

Research team: MBBS honours student from UNDA; research nurse; research academics; clinicians; statistician; pharmacist; secretarial support.

Equipment: Paper headache diary; NEC and sham drug capsules compounded by a pharmacy; computers; consulting space; telephone and website access; secure data base.

References available on request.

ELIGIBILITY:
Inclusion Criteria:

* Migraine (with or without aura) according to IHS 2013 criteria.

  * Migraine of at least one year's duration, with onset before 50 years of age.
  * Two-to-eight migraine episodes, and less than six 'other' headache types per month, averaged over 12 weeks prior to recruitment.
  * Subjects able to clearly distinguish between migraine and 'other' headache types.
  * Cognitive and English language skills allowing completion of headache diaries and self-administration of trial drugs.

Exclusion Criteria:

* Participation in a concurrent research trial.

  * Chronic daily headaches, according to IHS 2013 criteria.
  * Medication-overuse headache and/or other primary headache disorders, according to IHS 2013 criteria.
  * Change in migraine treatment in the twelve weeks prior to, or during the study.
  * Taking ≥ 2 migraine prevention drugs.
  * Failure to respond in ≥ 2 previous migraine prevention trials.
  * Taking NAc, VitE or VitC supplements in the 12 weeks prior to the study.
  * Pregnancy, or risk of pregnancy during the study; female of reproductive age not taking medically prescribed contraception; breast feeding.
  * Adverse reactions to NAc, VitE or VitC preparations; VitC deficiency.
  * Renal dysfunction (eGFR ≤ 30 ml/min/1.73m2), liver dysfunction (ALT or AST > 300 IU/L).
  * Clinical risks associated with bleeding, coagulopathy, warfarin therapy.
  * Haemochromatosis, glucose-6-phosphate dehydrogenase deficiency.
  * Daily opioid use in the 12 weeks prior to or during the study.
  * Substance abuse, dependence or addiction during the study.
  * Psychosis, bipolar affective disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Difference in mean number of migraine episodes per month between baseline and final four weeks of the study, for both study groups. | 16 weeks
  Difference in mean number of migraine episodes per month between baseline and final four weeks of the study, for both study groups.

SECONDARY OUTCOMES:
Difference in mean migraine duration (hours) per month between baseline and final four weeks of the study, for both study groups | 16 weeks
  Difference in mean migraine duration (hours) per month between baseline and final four weeks of the study, for both study groups
Difference in mean migraine severity score per month (categorical scale; 0 = nil, 1 = mild, 2 = moderate, 3 = severe) between baseline and final four weeks of the study, for both study groups. | 16 weeks
  Difference in mean migraine severity score per month (categorical scale; 0 = nil, 1 = mild, 2 = moderate, 3 = severe) between baseline and final four weeks of the study, for both study groups.
Difference in mean MIDAS per month between baseline and final four weeks of the study, for both study groups. | 16 weeks
  Migraine Disability Assessment Score (MIDAS).
Difference in mean MSQ score per month between baseline and final four weeks of the study, for both study groups. Migraine Specific Quality of Life Questionnaire (MSQ, Version 2.1) score. | 16 weeks
  Difference in mean MSQ score per month between baseline and final four weeks of the study, for both study groups. Migraine Specific Quality of Life Questionnaire (MSQ, Version 2.1) score.
Difference in mean HRQOL score per month between baseline and final four weeks of the study, for both study groups.Health Related Quality of Life (HRQOL) score | 16 weeks
  Difference in mean HRQOL score per month between baseline and final four weeks of the study, for both study groups.Health Related Quality of Life (HRQOL) score
Number of treatment adverse events per month Number and type of treatment-related adverse effects per month. Number and type of treatment-related adverse effect | 16 weeks
  Number of treatment adverse events per month
Difference in mean number of migraine days per month between baseline and final four weeks of the study, for both study groups. | 16 Weeks
  Difference in mean number of migraine days per month between baseline and final four weeks of the study, for both study groups.
Responder rate: Percentage of subjects reporting ≥ 30% reduction in migraine episodes per month between baseline and final four weeks of the study, for both study groups | 16 weeks
  Responder rate: Percentage of subjects reporting ≥ 30% reduction in migraine episodes per month between baseline and final four weeks of the study, for both study groups

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Visser, MBBS, Principal Investigator — University of Notre Dame Australia